CLINICAL TRIAL: NCT00853112
Title: A Phase 2a, Randomized, Double Blind, Placebo-controlled, Parallel Group Study Investigating The Dose-response Of Pf-00489791 On Acute Hemodynamics In Subjects With Idiopathic And Familial Pulmonary Arterial Hypertension
Brief Title: A Research Study To Assess The Effectiveness And Safety Of Different Doses Of Oral PF-00489791 In The Treatment Of Adult Patients With Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A7331009; 2008-003572-21 (EudraCT Number)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Hypertension, Pulmonary
Keywords: PAH pulmonary hypertension pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — PF-00489791; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- PF-00489791 1 mg (Experimental)
  Interventions: Drug: PF-00489791
- PF-00489791 2 mg (Experimental)
  Interventions: Drug: PF-00489791
- PF-00489791 4 mg (Experimental)
  Interventions: Drug: PF-00489791
- PF-00489791 10 mg (Experimental)
  Interventions: Drug: PF-00489791
- PF-00489791 20 mg (Experimental)
  Interventions: Drug: PF-00489791
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Sildenafil (Active Comparator): Observational comparator arm
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: PF-00489791 — tablet form, 1 mg, single dose (Day 1)
  Arms: PF-00489791 1 mg
Drug: PF-00489791 — tablet form, 2 mg, single dose (Day 1)
  Arms: PF-00489791 2 mg
Drug: PF-00489791 — tablet form, 4 mg, single dose (Day 1)
  Arms: PF-00489791 4 mg
Drug: PF-00489791 — tablet form, 10 mg, single dose (Day 1)
  Arms: PF-00489791 10 mg
Drug: PF-00489791 — tablet form, 20 mg, single dose (Day 1)
  Arms: PF-00489791 20 mg
Drug: placebo — tablet form, single dose (Day 1)
  Arms: Placebo
Drug: sildenafil — tablet form, 20 mg, single dose (Day 1)
  Other Names: Revatio
  Arms: Sildenafil

SUMMARY:
Study will assess PF-00489791 efficacy and safety in Pulmonary Arterial Hypertension (PAH)

DETAILED DESCRIPTION:
Pfizer decided to stop this trial early upon Stage 1 completion due to change in PF-00489791 development and not as a result of safety concerns for PF-00489791. Date of termination (LSLV) occurred on July 28, 2010.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic or familial pulmonary arterial hypertension (PAH)
* Mean PAP at least 25 mm Hg, PCWP < 15 mm Hg at rest
* For females of child-bearing potential negative pregnancy test at screening and use of contraception during the study and 4 weeks after its completion
* Signed and dated informed consent
* Willingness to comply with the study plan and procedures

Exclusion Criteria:

* pulmonary arterial hypertension (PAH)other than idiopathic or familial
* For females, pregnancy or lactation
* Use of specific PAH treatments, potent CYP3A4 inhibitors, protease inhibitors, alpha blockers or arginine 30 days prior tio randomization and during the study
* Change of dose or class of standard background PAH therapy, i.e. oxygen, calcium channel blockers, digoxin, diuretics 30 days prior tio randomization and during the study
* Large shift in altitude (defined as >5000 feet or 1524 meters) during 90 days prior to baseline visit and/or during the study visit
* Subjects with intracardiac shunts and/or serious heart, lung or other health conditions
* HIV positive subjects
* Subjects participating in another clinical trial with an investigational drug or device
* Subjects with degenerative retinal disorders, history of non-arteritic anterior ischemic optic neuropathy or untreated proliferative diabetic retinopathy
* Allergies and previous intolerance of PDE5 inhibitors
* Alcohol or drug abuse
* Blood donation during the study, or 1 month before or after the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (7):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - John C. Lincoln Hospital, North Mountain, Phoenix, Arizona
  - Shands at University of Florida, Gainesville, Florida
  - Creighton University Medical Center, Omaha, Nebraska
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center - Department of Internal Medicine Pulmonary, Dallas, Texas
  - UT Southwestern St. Paul Hospital, Dallas, Texas
- Canada (3):
  - Lawson Health Research Institute, London, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sir Mortimer B. Davis, Jewish General Hospital, Montreal, Quebec
- Thoraxklinik am Universitaetsklinikum, Heidelberg, Germany
- India (4):
  - Department Of Cardiology, MediCiti Hospital,, Hyderabad, Andhra Pardesh
  - Department Of Cardiology, Sri Venkateswara Institute Of Medical Sciences, Tirupati, Andhra Pardesh
  - Bankers Heart Institute, Vadodara, Gujarat
  - Omega Hospital, Mangalore, Karnataka
- Russia (2):
  - Moscow Healthcare Institution "City Clinical Hospital No. 57", Moscow
  - Institute of Cardiosurgery n.a. V.I.Burakovsky, Moscow
- Spain (3):
  - Hospital General Universitari Vall D´Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (3):
  - Universitetssjukhuset i Lund, Hjart- och Lungdivisionen, Lund
  - Norrlands Universitetssjukhus, Kliniskt Forsknings Centrum, Umeå
  - Akademiska Sjukhuset, Kardiologen 50F/Forskningsenheten, Uppsala
- Universitaetsspittal Zuerich, Medizinische Klinik A, Zurich, Switzerland

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7331009&StudyName=A%20Research%20Study%20To%20Assess%20The%20Effectiveness%20And%20Safety%20Of%20Different%20Doses%20Of%20Oral%20PF-00489791%20In%20The%20Treatment%20Of%20Adult%20Patients%20Wi

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single oral dose of 2 placebo matched to PF-00489791 tablet along with 1 placebo matched to sildenafil tablet on Day 1.
- PF-00489791 1 mg: Single oral dose of 1 PF-00489791 1 milligram (mg) tablet along with 1 placebo matched to PF-00489791 tablet and 1 placebo matched to sildenafil tablet on Day 1.
- PF-00489791 2 mg: Single oral dose of 1 PF-00489791 2 mg tablet along with 1 placebo matched to PF-00489791 tablet and 1 placebo matched to sildenafil tablet on Day 1.
- PF-00489791 4 mg: Single oral dose of 2 PF-00489791 2 mg tablet (equivalent to PF-00489791 4 mg) along with 1 placebo matched to sildenafil tablet on Day 1.
- PF-00489791 10 mg: Single oral dose of 1 PF-00489791 10 mg tablet along with 1 placebo matched to PF-00489791 tablet and 1 placebo matched to sildenafil tablet on Day 1.
- PF-00489791 20 mg: Single oral dose of 2 PF-00489791 10 mg tablet (equivalent to PF-00489791 20 mg) along with 1 placebo matched to sildenafil tablet on Day 1.
- Sildenafil: Single oral dose of 1 sildenafil 20 mg tablet along with 2 placebo matched to PF-00489791 tablet on Day 1.
Period: Overall Study
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Started | 6 | 7 | 7 | 8 | 6 | 7 | 7
Treated | 6 | 6 | 7 | 6 | 6 | 7 | 6
Completed | 6 | 6 | 7 | 6 | 6 | 7 | 6
Not Completed | 0 | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Randomized but not treated | 0 | 1 | 0 | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6 | 44
Age, Customized [Number; unit: participants]
  Between 18 and 44 Years | 3 | 2 | 4 | 5 | 2 | 2 | 3 | 21
  Between 45 and 64 Years | 2 | 1 | 3 | 0 | 2 | 3 | 2 | 13
  Greater than or equal to (>=) 65 Years | 1 | 3 | 0 | 1 | 2 | 2 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 4 | 3 | 5 | 4 | 30
  Male | 1 | 1 | 3 | 2 | 3 | 2 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Pulmonary Vascular Resistance Index (PVRI) Over 4 Hours Post Dose
Description: PVRI was calculated as: PVRI (in Wood units*meter^2 [m^2]) = pulmonary vascular resistance (PVR) multiplied by body surface area (BSA). PVR (in Wood units) = (mean pulmonary artery pressure [mean PAP] minus pulmonary capillary wedge pressure [PCWP]) divided by cardiac output (CO, taken as the average of the triplicate measurements). BSA (m^2) = (0.007184) multiplied by (height in centimeters [cm])^0.725 multiplied by (weight in kilograms [kg])^0.425. PVRI values were converted to dyne*second (s)*m^2/centimeter (cm)^5 from Woods units by multiplying by a factor of 79.9. The change from baseline in PVRI over 4-hour interval was calculated as the average of the change from baseline values at 1, 2, 3, and 4 hours post dose on Day 1.
Time Frame: Baseline, up to 4 hours post-dose on Day 1
Population: Full analysis set (FAS) included all randomized participants who received study medication. Here, N (overall number of participants analyzed) = participants evaluable for this measure and 'Number Analyzed' = participants who were evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: (dyne*s*m^2)/cm^5
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
(dyne*s*m^2)/cm^5
  Baseline | 2026.5 (1141.94) | 1043.1 (327.07) | 1602.4 (990.36) | 1934.3 (675.31) | 1328.2 (784.24) | 1380.8 (1058.35) | 1674.0 (925.53)
  Change over 4 hours post-dose: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 5 | 5
  Change over 4 hours post-dose | -47.3 (507.90) | -106.8 (136.41) | 11.6 (213.55) | -335.3 (499.52) | -267.0 (397.56) | -254.0 (361.07) | 304.9 (799.78)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; Change over 4 hours post-dose: The Bayesian 4-parameter Emax model was used for analysis. 95% credible intervals of the effect size and the posterior distribution were calculated. Posterior distribution was used to calculate a probability (presented as p value) that the dose gives a difference of >=240 dyne*s*m^2/cm^5 from placebo. The predicted means and SD were the posterior means and standard deviation (SD) from the Bayesian analysis; Test type: Superiority or Other; p = 0.120, Bayesian 4-parameter Emax model; Predicted Mean Difference = -115.0, 95% CI 2-sided [-371.5 to -1.1], Standard Deviation 98.36
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; Change over 4 hours post-dose: The Bayesian 4-parameter Emax model was used for analysis. 95% credible intervals of the effect size and the posterior distribution were calculated. Posterior distribution was used to calculate a probability (presented as p value) that the dose gives a difference of >=240 dyne.s.m2/cm5 from placebo. The predicted means and SD were the posterior means and SD from the Bayesian analysis; Test type: Superiority or Other; p = 0.250, Bayesian 4-parameter Emax model; Predicted Mean Difference = -170.6, 95% CI 2-sided [-409.2 to -7.1], Standard Deviation 107.84
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; The Bayesian 4-parameter Emax model was used for analysis. 95% credible intervals of the effect size and the posterior distribution were calculated. Posterior distribution was used to calculate a probability (presented as p value) that the dose gives a difference of >=240 dyne*s*m^2/cm^5 from placebo. The predicted means and SD were the posterior means and SD from the Bayesian analysis; Test type: Superiority or Other; p = 0.485, Bayesian 4-parameter Emax model; Predicted Mean Difference = -240.2, 95% CI 2-sided [-444.8 to -33.8], Standard Deviation 109.28
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; Change over 4 hours post-dose: The Bayesian 4-parameter Emax model was used for analysis. 95% credible intervals of the effect size and the posterior distribution were calculated. Posterior distribution was used to calculate a probability (presented as p value) that the dose gives a difference of >=240 dyne*s*m^2/cm^5 from placebo. The predicted means and SD were the posterior means and SD from the Bayesian analysis; Test type: Superiority or Other; p = 0.810, Bayesian 4-parameter Emax model; Predicted Mean Difference = -327.9, 95% CI 2-sided [-492.9 to -148.0], Standard Deviation 92.41
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; Change over 4 hours post-dose: The Bayesian 4-parameter Emax model was used for analysis. Posterior distribution was calculated and was used to calculate a probability (presented as p value) that the dose gives a difference of >=240 dyne*s*m^2/cm^5 from placebo. The predicted means and SD were the posterior means and SD from the Bayesian analysis; Test type: Superiority or Other; p = 0.974, Bayesian 4-parameter Emax model; Predicted Mean Difference = -379.4, 95% CI 2-sided [-520.6 to -238.8], Standard Deviation 73.61

2. Secondary Outcome: Greatest Reduction From Baseline in Pulmonary Vascular Resistance Index (PVRI) and Systemic Vascular Resistance Index (SVRI) Over 4 Hours Post Dose
Description: PVRI was calculated as: PVRI (in Wood units*m^2) = PVR multiplied by BSA. PVR (in Wood units) = (mean PAP minus PCWP) divided by CO (taken as the average of the triplicate measurements). SVRI was calculated as: SVRI (Wood units*m^2) = systemic vascular resistance (SVR) multiplied by BSA. SVR (Wood units) = (mean systemic arterial pressure [mean SAP] minus right atrial pressure [RAP]) divided by CO (taken as the average of the triplicate measurements). BSA (m^2) = (0.007184) multiplied by (height in cm)^0.725 multiplied by (weight in kg)^0.425. PVRI and SVRI values were converted to dyne*s*m^2/cm^5 from Woods units by multiplying by a factor of 79.9. For each participant the greatest reduction (GR) from baseline in PVRI and SVRI over 4-hour interval was defined as the maximum reduction (greatest decrease or smallest increase) observed at 1, 2, 3, and 4 hours post dose on Day 1.
Time Frame: Baseline, up to 4 hours post-dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (dyne*s*m^2)/cm^5
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
(dyne*s*m^2)/cm^5
  Baseline: SVRI | 3560.6 (1481.67) | 2512.2 (858.62) | 2599.6 (874.85) | 3679.1 (1248.03) | 3175.8 (644.80) | 2577.1 (791.93) | 3121.8 (544.52)
  GR over 4 hours: PVRI: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 5 | 5
  GR over 4 hours: PVRI | -180.8 (487.37) | -210.2 (132.60) | -143.4 (188.58) | -600.9 (453.38) | -397.8 (386.51) | -385.9 (455.07) | 55.8 (526.85)
  GR over 4 hours: SVRI | -806.1 (480.86) | -387.6 (428.39) | -394.1 (594.61) | -1110.5 (1079.75) | -1000.6 (529.43) | -524.1 (370.71) | -113.6 (726.61)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; GR over 4 hours, PVRI: The analysis was performed using Analysis of Covariance (ANCOVA) with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.354, ANCOVA; Adjusted Mean Difference = -195.3, 95% CI 2-sided [-618.8 to 228.3], Standard Error of Mean 207.38
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; GR over 4 hours, PVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.860, ANCOVA; Adjusted Mean Difference = -34.1, 95% CI 2-sided [-424.1 to 356.0], Standard Error of Mean 190.99
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; GR over 4 hours, PVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.034, ANCOVA; Adjusted Mean Difference = -435.7, 95% CI 2-sided [-835.9 to -35.6], Standard Error of Mean 195.94
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; GR over 4 hours, PVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.107, ANCOVA; Adjusted Mean Difference = -334.7, 95% CI 2-sided [-746.7 to 77.3], Standard Error of Mean 201.74
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; GR over 4 hours, PVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.177, ANCOVA; Adjusted Mean Difference = -278.0, 95% CI 2-sided [-688.3 to 132.2], Standard Error of Mean 200.89
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 1 mg; GR over 4 hours, SVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.873, ANCOVA; Mean Difference (Final Values) = 51.1, 95% CI 2-sided [-594.1 to 696.3], Standard Error of Mean 315.91
Statistical Analysis 7: Comparison: Placebo vs PF-00489791 2 mg; GR over 4 hours, SVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.806, ANCOVA; Adjusted Mean Difference = 75.2, 95% CI 2-sided [-543.8 to 694.1], Standard Error of Mean 303.08
Statistical Analysis 8: Comparison: Placebo vs PF-00489791 4 mg; GR over 4 hours, SVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.390, ANCOVA; Adjusted Mean Difference = -262.8, 95% CI 2-sided [-877.8 to 352.1], Standard Error of Mean 301.10
Statistical Analysis 9: Comparison: Placebo vs PF-00489791 10 mg; GR over 4 hours, SVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.286, ANCOVA; Adjusted Mean Difference = -329.4, 95% CI 2-sided [-948.1 to 289.4], Standard Error of Mean 302.97
Statistical Analysis 10: Comparison: Placebo vs PF-00489791 20 mg; GR over 4 hours, SVRI: The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.843, ANCOVA; Adjusted Mean Difference = -62.7, 95% CI 2-sided [-704.3 to 578.9], Standard Error of Mean 314.15

3. Secondary Outcome: Mean Change From Baseline in Systemic Vascular Resistance Index (SVRI) Over 4 Hours Post Dose
Description: SVRI was calculated as: SVRI (Wood units*m^2) = SVR multiplied by BSA. SVR (Wood units) = (mean SAP minus RAP) divided by CO (taken as the average of the triplicate measurements). BSA (m^2) = (0.007184) multiplied by (height in cm)^0.725 multiplied by (weight in kg)^0.425. SVRI values were converted to dyne*s*m^2/cm^5 from Woods units by multiplying by a factor of 79.9. The change from baseline in SVRI over 4-hour interval was calculated as the average of the change from baseline values at 1, 2, 3, and 4 hours post dose on Day 1.
Time Frame: Baseline, up to 4 hours post-dose on Day 1
Population: FAS included all randomized participants who received study medication. Here, N (overall number of participants analyzed) = participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: (dyne*s*m^2)/cm^5
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
(dyne*s*m^2)/cm^5 | -486.8 (543.83) | -193.9 (336.10) | -145.7 (557.67) | -609.6 (1061.78) | -704.7 (501.01) | -272.8 (228.53) | 97.6 (810.82)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.999, ANCOVA; Adjusted Mean Difference = -0.4, 95% CI 2-sided [-659.7 to 658.8], Standard Error of Mean 322.80
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.817, ANCOVA; Adjusted Mean Difference = 72.2, 95% CI 2-sided [-560.2 to 704.7], Standard Error of Mean 309.69
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.790, ANCOVA; Adjusted Mean Difference = -82.6, 95% CI 2-sided [-711.0 to 545.7], Standard Error of Mean 307.67
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.301, ANCOVA; Adjusted Mean Difference = -325.6, 95% CI 2-sided [-957.8 to 306.7], Standard Error of Mean 309.58
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; The analysis was performed using ANCOVA with baseline fitted as a covariate; Test type: Superiority or Other; p = 0.850, ANCOVA; Adjusted Mean Difference = -61.2, 95% CI 2-sided [-716.8 to 594.4], Standard Error of Mean 321.00

4. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance Index (PVRI) at Hour 1, 2, 3 and 4 Post Dose
Description: PVRI was calculated as: PVR multiplied by BSA. PVR = (mean PAP minus PCWP) divided by CO (taken as the average of the triplicate measurements). BSA (m^2) = 0.007184 times height (cm)^0.725 times weight (kilogram)^0.425. Wood unit equals to 79.9 dyne*second/cm^5. Hourly changes from baseline in PVRI was reported.
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: FAS included all randomized participants who received study medication. Here, N (overall number of participants analyzed) = participants evaluable for this measure and 'Number Analyzed' = participants who were evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: (dyne*s*m^2)/cm^5
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
(dyne*s*m^2)/cm^5
  Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 5 | 5
  Change at hour 1 | 32.03 (637.84) | -121.86 (228.17) | -15.84 (245.75) | -333.75 (482.43) | -228.30 (526.40) | -183.51 (123.88) | 121.33 (449.03)
  Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 4 | 6 | 5 | 5
  Change at hour 2 | -84.78 (554.32) | -167.42 (169.75) | 2.91 (216.15) | -210.86 (779.62) | -302.42 (378.43) | -315.71 (441.19) | 252.41 (891.95)
  Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 4 | 6 | 5 | 5
  Change at hour 3 | -51.15 (501.81) | -22.45 (182.54) | 16.64 (272.36) | -326.88 (815.60) | -244.54 (367.99) | -276.37 (519.49) | 392.24 (859.17)
  Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 5 | 5
  Change at hour 4 | -85.20 (406.10) | -115.49 (172.46) | 42.55 (321.24) | -416.28 (420.63) | -292.65 (399.71) | -240.48 (422.15) | 453.54 (1012.97)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.295, Longitudinal analysis; Adjusted Mean Difference = -269.32, 95% CI 2-sided [-785.39 to 246.76], Standard Error of Mean 252.93
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.680, Longitudinal analysis; Adjusted Mean Difference = -97.65, 95% CI 2-sided [-577.02 to 381.72], Standard Error of Mean 234.55
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.129, Longitudinal analysis; Adjusted Mean Difference = -376.61, 95% CI 2-sided [-869.53 to 116.31], Standard Error of Mean 241.06
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.176, Longitudinal analysis; Adjusted Mean Difference = -342.29, 95% CI 2-sided [-846.90 to 162.32], Standard Error of Mean 247.07
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; Hour 1: Longitudinal analysis was used to analyze p-value and included baseline as a covariate; Test type: Superiority or Other; p = 0.235, Longitudinal analysis; Mean Difference (Final Values) = -316.86, 95% CI 2-sided [-850.90 to 217.17], Standard Error of Mean 261.58
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.430, Longitudinal analysis; Adjusted Mean Difference = -198.06, 95% CI 2-sided [-705.04 to 308.91], Standard Error of Mean 247.62
Statistical Analysis 7: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.870, Longitudinal analysis; Adjusted Mean Difference = 37.90, 95% CI 2-sided [-432.23 to 508.04], Standard Error of Mean 229.23
Statistical Analysis 8: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.645, Longitudinal analysis; Adjusted Mean Difference = -114.06, 95% CI 2-sided [-614.57 to 386.45], Standard Error of Mean 244.95
Statistical Analysis 9: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.225, Longitudinal analysis; Adjusted Mean Difference = -299.60, 95% CI 2-sided [-794.81 to 195.61], Standard Error of Mean 241.63
Statistical Analysis 10: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.205, Longitudinal analysis; Adjusted Mean Difference = -332.25, 95% CI 2-sided [-856.55 to 192.05], Standard Error of Mean 255.93
Statistical Analysis 11: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.745, Longitudinal analysis; Adjusted Mean Difference = -86.72, 95% CI 2-sided [-625.87 to 452.42], Standard Error of Mean 263.63
Statistical Analysis 12: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.942, Longitudinal analysis; Adjusted Mean Difference = 18.00, 95% CI 2-sided [-484.46 to 520.47], Standard Error of Mean 245.25
Statistical Analysis 13: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.314, Longitudinal analysis; Adjusted Mean Difference = -265.94, 95% CI 2-sided [-796.15 to 264.28], Standard Error of Mean 259.53
Statistical Analysis 14: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.295, Longitudinal analysis; Adjusted Mean Difference = -275.35, 95% CI 2-sided [-803.57 to 252.88], Standard Error of Mean 258.01
Statistical Analysis 15: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.241, Longitudinal analysis; Adjusted Mean Difference = -326.55, 95% CI 2-sided [-885.12 to 232.02], Standard Error of Mean 272.96
Statistical Analysis 16: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.510, Longitudinal analysis; Adjusted Mean Difference = -145.71, 95% CI 2-sided [-592.24 to 300.83], Standard Error of Mean 218.50
Statistical Analysis 17: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.699, Longitudinal analysis; Adjusted Mean Difference = 77.96, 95% CI 2-sided [-330.70 to 486.63], Standard Error of Mean 199.85
Statistical Analysis 18: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.106, Longitudinal analysis; Adjusted Mean Difference = -341.91, 95% CI 2-sided [-760.45 to 76.64], Standard Error of Mean 204.65
Statistical Analysis 19: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.182, Longitudinal analysis; Adjusted Mean Difference = -289.41, 95% CI 2-sided [-722.17 to 143.35], Standard Error of Mean 211.69
Statistical Analysis 20: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.263, Longitudinal analysis; Adjusted Mean Difference = -256.60, 95% CI 2-sided [-716.26 to 203.06], Standard Error of Mean 224.88

5. Secondary Outcome: Change From Baseline in Systemic Vascular Resistance Index (SVRI) at Hour 1, 2, 3 and 4 Post Dose
Description: SVRI is the product of SVR and BSA. SVR equals to (mean SAP subtracted by RAP) divided by CO (taken as the average of the triplicate measurements). BSA (m^2) equals to 0.007184 times height (cm)^0.725 times weight (kilogram) ^0.425. Wood unit equals to 79.9 dyne*second/cm^5. Hourly changes from baseline in SVRI was reported.
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: (dyne*s*m^2)/cm^5
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
(dyne*s*m^2)/cm^5
  Change at hour 1 | -278.74 (812.16) | -281.26 (386.52) | -145.25 (712.56) | -602.63 (993.10) | -616.40 (674.29) | -48.54 (218.85) | 125.71 (607.77)
  Change at hour 2 | -518.41 (533.85) | -308.47 (487.47) | -222.83 (550.92) | -381.01 (1069.58) | -893.81 (479.01) | -347.45 (392.26) | 34.44 (959.10)
  Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 5 | 6 | 6 | 6
  Change at hour 3 | -489.10 (531.15) | -115.91 (321.47) | -92.23 (551.76) | -502.93 (1390.25) | -739.16 (485.07) | -369.29 (423.35) | 79.04 (844.22)
  Change at hour 4 | -660.98 (524.55) | -69.89 (290.88) | -122.36 (560.20) | -874.51 (1171.91) | -569.43 (581.07) | -325.95 (372.51) | 151.18 (902.51)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.401, Longitudinal analysis; Adjusted Mean Difference = -328.10, 95% CI 2-sided [-1114.11 to 457.92], Standard Error of Mean 385.78
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.659, Longitudinal analysis; Adjusted Mean Difference = -164.96, 95% CI 2-sided [-920.05 to 590.12], Standard Error of Mean 370.54
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.447, Longitudinal analysis; Adjusted Mean Difference = -287.08, 95% CI 2-sided [-1047.59 to 473.42], Standard Error of Mean 372.60
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.231, Longitudinal analysis; Adjusted Mean Difference = -457.16, 95% CI 2-sided [-1220.86 to 306.53], Standard Error of Mean 374.26
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.846, Longitudinal analysis; Adjusted Mean Difference = -75.24, 95% CI 2-sided [-858.19 to 707.71], Standard Error of Mean 384.20
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.748, Longitudinal analysis; Adjusted Mean Difference = -115.64, 95% CI 2-sided [-844.24 to 612.96], Standard Error of Mean 357.20
Statistical Analysis 7: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.993, Longitudinal analysis; Adjusted Mean Difference = -2.87, 95% CI 2-sided [-702.41 to 696.67], Standard Error of Mean 342.91
Statistical Analysis 8: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.615, Longitudinal analysis; Adjusted Mean Difference = 174.20, 95% CI 2-sided [-526.41 to 874.81], Standard Error of Mean 342.93
Statistical Analysis 9: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.161, Longitudinal analysis; Adjusted Mean Difference = -494.91, 95% CI 2-sided [-1199.04 to 209.21], Standard Error of Mean 344.72
Statistical Analysis 10: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.708, Longitudinal analysis; Adjusted Mean Difference = -134.48, 95% CI 2-sided [-859.74 to 590.77], Standard Error of Mean 355.50
Statistical Analysis 11: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.897, Longitudinal analysis; Adjusted Mean Difference = 47.61, 95% CI 2-sided [-697.56 to 792.79], Standard Error of Mean 365.43
Statistical Analysis 12: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.781, Longitudinal analysis; Adjusted Mean Difference = 98.42, 95% CI 2-sided [-617.15 to 813.99], Standard Error of Mean 350.87
Statistical Analysis 13: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.937, Longitudinal analysis; Adjusted Mean Difference = -28.31, 95% CI 2-sided [-753.46 to 696.83], Standard Error of Mean 355.47
Statistical Analysis 14: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.304, Longitudinal analysis; Adjusted Mean Difference = -369.57, 95% CI 2-sided [-1090.86 to 351.72], Standard Error of Mean 353.25
Statistical Analysis 15: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.613, Longitudinal analysis; Adjusted Mean Difference = -185.64, 95% CI 2-sided [-927.54 to 556.27], Standard Error of Mean 363.77
Statistical Analysis 16: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.420, Longitudinal analysis; Adjusted Mean Difference = 265.51, 95% CI 2-sided [-397.45 to 928.48], Standard Error of Mean 324.88
Statistical Analysis 17: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.447, Longitudinal analysis; Adjusted Mean Difference = 240.17, 95% CI 2-sided [-395.81 to 876.14], Standard Error of Mean 311.63
Statistical Analysis 18: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.572, Longitudinal analysis; Adjusted Mean Difference = -176.74, 95% CI 2-sided [-808.10 to 454.63], Standard Error of Mean 309.11
Statistical Analysis 19: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.929, Longitudinal analysis; Adjusted Mean Difference = -27.96, 95% CI 2-sided [-663.31 to 607.38], Standard Error of Mean 311.11
Statistical Analysis 20: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.928, Longitudinal analysis; Adjusted Mean Difference = 29.58, 95% CI 2-sided [-629.62 to 688.79], Standard Error of Mean 323.01

6. Secondary Outcome: Change From Baseline in Cardiac Index (CI) at Hour 1, 2, 3 and 4 Post Dose
Description: CI was calculated as: CI (liters per minute per square meter [L/min/m^2]) = CO (taken as the average of the triplicate measurements) divided by BSA. BSA (m^2) = (0.007184) multiplied by (height in cm)^0.725 multiplied by (weight in kg)^0.425.
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
L/min/m^2
  Baseline | 1.90 (0.50) | 2.90 (0.69) | 2.99 (1.61) | 2.05 (0.55) | 2.30 (0.40) | 3.07 (1.47) | 2.43 (0.70)
  Change at hour 1 | 0.12 (0.25) | 0.20 (0.57) | -0.06 (0.67) | 0.27 (0.36) | 0.49 (0.67) | -0.13 (0.21) | -0.15 (0.31)
  Change at hour 2 | 0.22 (0.24) | 0.36 (0.78) | 0.09 (0.65) | 0.17 (0.46) | 0.59 (0.41) | 0.14 (0.88) | -0.11 (0.45)
  Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 5 | 6 | 6 | 6
  Change at hour 3 | 0.19 (0.29) | 0.12 (0.31) | -0.15 (0.77) | 0.19 (0.41) | 0.54 (0.62) | 0.19 (0.63) | -0.24 (0.26)
  Change at hour 4 | 0.20 (0.36) | 0.10 (0.56) | -0.12 (0.59) | 0.36 (0.30) | 0.38 (0.54) | 0.26 (0.38) | -0.27 (0.29)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.412, Longitudinal analysis; Adjusted Mean Difference = 0.24, 95% CI 2-sided [-0.35 to 0.83], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.999, Longitudinal analysis; Adjusted Mean Difference = 0.00, 95% CI 2-sided [-0.58 to 0.58], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.535, Longitudinal analysis; Adjusted Mean Difference = 0.17, 95% CI 2-sided [-0.39 to 0.74], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.128, Longitudinal analysis; Adjusted Mean Difference = 0.44, 95% CI 2-sided [-0.13 to 1.01], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.823, Longitudinal analysis; Adjusted Mean Difference = -0.07, 95% CI 2-sided [-0.67 to 0.53], Standard Error of Mean 0.29
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.396, Longitudinal analysis; Adjusted Mean Difference = 0.29, 95% CI 2-sided [-0.40 to 0.99], Standard Error of Mean 0.34
Statistical Analysis 7: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.899, Longitudinal analysis; Adjusted Mean Difference = 0.04, 95% CI 2-sided [-0.63 to 0.72], Standard Error of Mean 0.33
Statistical Analysis 8: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.928, Longitudinal analysis; Adjusted Mean Difference = -0.03, 95% CI 2-sided [-0.70 to 0.64], Standard Error of Mean 0.33
Statistical Analysis 9: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.203, Longitudinal analysis; Adjusted Mean Difference = 0.43, 95% CI 2-sided [-0.25 to 1.11], Standard Error of Mean 0.33
Statistical Analysis 10: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.772, Longitudinal analysis; Adjusted Mean Difference = 0.10, 95% CI 2-sided [-0.60 to 0.80], Standard Error of Mean 0.34
Statistical Analysis 11: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.771, Longitudinal analysis; Adjusted Mean Difference = 0.09, 95% CI 2-sided [-0.52 to 0.69], Standard Error of Mean 0.29
Statistical Analysis 12: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.572, Longitudinal analysis; Adjusted Mean Difference = -0.16, 95% CI 2-sided [-0.75 to 0.42], Standard Error of Mean 0.29
Statistical Analysis 13: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.966, Longitudinal analysis; Adjusted Mean Difference = 0.01, 95% CI 2-sided [-0.58 to 0.60], Standard Error of Mean 0.29
Statistical Analysis 14: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.157, Longitudinal analysis; Adjusted Mean Difference = 0.41, 95% CI 2-sided [-0.17 to 1.00], Standard Error of Mean 0.28
Statistical Analysis 15: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.546, Longitudinal analysis; Adjusted Mean Difference = 0.18, 95% CI 2-sided [-0.43 to 0.79], Standard Error of Mean 0.30
Statistical Analysis 16: Comparison: Placebo vs PF-00489791 1 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.818, Longitudinal analysis; Adjusted Mean Difference = 0.07, 95% CI 2-sided [-0.51 to 0.64], Standard Error of Mean 0.28
Statistical Analysis 17: Comparison: Placebo vs PF-00489791 2 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.603, Longitudinal analysis; Adjusted Mean Difference = -0.14, 95% CI 2-sided [-0.71 to 0.42], Standard Error of Mean 0.28
Statistical Analysis 18: Comparison: Placebo vs PF-00489791 4 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.495, Longitudinal analysis; Adjusted Mean Difference = 0.19, 95% CI 2-sided [-0.37 to 0.74], Standard Error of Mean 0.27
Statistical Analysis 19: Comparison: Placebo vs PF-00489791 10 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.375, Longitudinal analysis; Adjusted Mean Difference = 0.24, 95% CI 2-sided [-0.31 to 0.80], Standard Error of Mean 0.27
Statistical Analysis 20: Comparison: Placebo vs PF-00489791 20 mg; Change at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.392, Longitudinal analysis; Adjusted Mean Difference = 0.25, 95% CI 2-sided [-0.34 to 0.84], Standard Error of Mean 0.29

7. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (mPAP), Systolic Pulmonary Artery Pressure (sPAP), Diastolic Pulmonary Artery Pressure (dPAP), Right Atrial Pressure (RAP) at Hour 1, 2, 3 and 4 Post Dose
Description: Hourly changes from baseline in hemodynamic parameters were reported. Hemodynamic parameters including mPAP, sPAP, dPAP and RAP were measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position. All hemodynamic pressure measurements were performed as triplicate measurements and average was used.
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: FAS included all randomized participants who received study medication. Here, 'Number Analyzed' = participants who were evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6
millimeters of mercury (mmHg)
  Baseline: mPAP: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  Baseline: mPAP | 53.67 (15.36) | 45.67 (13.47) | 60.29 (22.32) | 53.83 (11.34) | 44.95 (18.98) | 50.17 (23.25) | 55.33 (18.49)
  Baseline: sPAP | 88.3 (20.69) | 71.2 (17.84) | 84.1 (32.62) | 83.8 (24.26) | 68.2 (28.93) | 68.6 (29.53) | 82.5 (28.13)
  Baseline: dPAP | 34.5 (13.28) | 29.3 (12.86) | 45.0 (17.51) | 35.7 (8.71) | 29.7 (14.68) | 39.1 (18.41) | 41.0 (16.63)
  Baseline: RAP | 11.5 (5.01) | 5.3 (3.72) | 9.3 (2.21) | 8.5 (4.32) | 5.7 (1.37) | 8.3 (3.64) | 6.5 (3.27)
  mPAP: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  mPAP: Change at hour 1 | 2.17 (8.89) | -3.00 (4.47) | -2.00 (5.23) | -1.50 (7.69) | 0.38 (6.23) | -6.00 (4.43) | -2.67 (6.92)
  sPAP: Change at hour 1 | 1.0 (13.96) | -5.3 (5.79) | -3.3 (6.52) | -3.0 (13.19) | -2.8 (10.34) | -7.0 (8.21) | -6.5 (11.15)
  dPAP: Change at hour 1 | 2.2 (6.68) | -0.3 (5.09) | -2.3 (4.61) | -0.5 (6.72) | 4.7 (6.59) | -6.4 (5.86) | -2.0 (3.03)
  RAP: Change at hour 1 | 0.3 (1.03) | 1.2 (1.47) | -1.0 (1.83) | -1.3 (2.73) | 0.2 (1.47) | -1.4 (2.99) | -0.3 (1.37)
  mPAP: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  mPAP: Change at hour 2 | 2.83 (7.17) | -3.67 (4.72) | 1.29 (5.74) | -0.83 (6.77) | 1.05 (5.12) | -5.50 (4.14) | -1.00 (6.07)
  sPAP: Change at hour 2 | 8.3 (13.47) | -8.5 (8.92) | -0.6 (8.92) | -4.2 (11.46) | -1.7 (7.92) | -6.4 (7.37) | -6.5 (8.19)
  dPAP: Change at hour 2 | 0.7 (3.50) | -0.5 (7.34) | 1.6 (4.65) | -0.5 (7.26) | 3.8 (6.05) | -7.3 (3.55) | -0.3 (3.61)
  RAP: Change at hour 2 | 1.0 (1.55) | 0.0 (1.10) | -1.0 (1.83) | -1.5 (1.87) | 0.5 (1.76) | -1.0 (2.52) | 0.0 (1.90)
  mPAP: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  mPAP: Change at hour 3 | 2.83 (5.27) | 1.17 (7.94) | -1.71 (7.80) | -3.17 (3.87) | 2.10 (6.64) | -6.33 (5.96) | -0.67 (7.50)
  sPAP: Change at hour 3 | 5.0 (5.83) | -2.8 (7.63) | -5.0 (10.88) | -4.0 (10.83) | -1.3 (10.35) | -8.6 (10.49) | -4.5 (8.92)
  dPAP: Change at hour 3 | 1.7 (6.53) | 3.3 (10.60) | -0.4 (5.50) | -1.8 (4.49) | 4.8 (9.11) | -6.7 (5.44) | -1.3 (2.94)
  RAP: Change at hour 3 | 1.3 (3.01) | 0.5 (1.38) | -1.1 (2.27) | 0.8 (5.04) | 0.7 (2.25) | -2.4 (3.51) | -0.2 (1.72)
  mPAP: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  mPAP: Change at hour 4 | 2.67 (6.47) | -3.50 (5.54) | -0.86 (9.32) | -2.50 (2.74) | -0.28 (6.48) | -6.33 (6.53) | -0.67 (9.03)
  sPAP: Change at hour 4 | 0.3 (11.91) | -7.7 (10.56) | -4.9 (14.42) | -3.3 (10.23) | -8.7 (8.76) | -4.9 (11.58) | -3.7 (11.60)
  dPAP: Change at hour 4 | 3.7 (6.77) | -0.7 (5.54) | 1.1 (7.03) | -2.2 (4.36) | 5.3 (8.26) | -8.9 (8.59) | -1.0 (4.20)
  RAP: Change at hour 4 | 1.2 (2.71) | 1.0 (2.00) | -0.7 (2.56) | 0.0 (4.60) | 0.3 (2.42) | -1.7 (3.09) | 0.5 (3.33)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 1 mg; mPAP at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.210, Longitudinal analysis; Adjusted Mean Difference = -4.80, 95% CI 2-sided [-12.47 to 2.86], Standard Error of Mean 3.75
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 2 mg; mPAP at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.225, Longitudinal analysis; Adjusted Mean Difference = -4.47, 95% CI 2-sided [-11.84 to 2.90], Standard Error of Mean 3.61
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 4 mg; mPAP at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.332, Longitudinal analysis; Adjusted Mean Difference = -3.67, 95% CI 2-sided [-11.28 to 3.93], Standard Error of Mean 3.73
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 10 mg; mPAP at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.714, Longitudinal analysis; Adjusted Mean Difference = -1.39, 95% CI 2-sided [-9.06 to 6.28], Standard Error of Mean 3.76
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 20 mg; mPAP at Hour 1: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.040, Longitudinal analysis; Adjusted Mean Difference = -8.01, 95% CI 2-sided [-15.63 to -0.39], Standard Error of Mean 3.73
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 1 mg; mPAP at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.079, Longitudinal analysis; Adjusted Mean Difference = -6.14, 95% CI 2-sided [-13.02 to 0.75], Standard Error of Mean 3.37
Statistical Analysis 7: Comparison: Placebo vs PF-00489791 2 mg; mPAP at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.573, Longitudinal analysis; Adjusted Mean Difference = -1.85, 95% CI 2-sided [-8.46 to 4.77], Standard Error of Mean 3.24
Statistical Analysis 8: Comparison: Placebo vs PF-00489791 4 mg; mPAP at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.280, Longitudinal analysis; Adjusted Mean Difference = -3.67, 95% CI 2-sided [-10.50 to 3.15], Standard Error of Mean 3.34
Statistical Analysis 9: Comparison: Placebo vs PF-00489791 10 mg; mPAP at Hour 2: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.684, Longitudinal analysis; Adjusted Mean Difference = -1.39, 95% CI 2-sided [-8.28 to 5.51], Standard Error of Mean 3.38
Statistical Analysis 10: Comparison: Placebo vs PF-00489791 20 mg; mPAP at Hour 2: Longitudinal analysis was used to analyze p-value and included baseline as a covariate; Test type: Superiority or Other; p = 0.021, Longitudinal analysis; Mean Difference (Final Values) = -8.17, 95% CI 2-sided [-15.01 to -1.34], Standard Error of Mean 3.35
Statistical Analysis 11: Comparison: Placebo vs PF-00489791 1 mg; mPAP at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.727, Longitudinal analysis; Adjusted Mean Difference = -1.30, 95% CI 2-sided [-8.86 to 6.25], Standard Error of Mean 3.70
Statistical Analysis 12: Comparison: Placebo vs PF-00489791 2 mg; mPAP at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.183, Longitudinal analysis; Adjusted Mean Difference = -4.85, 95% CI 2-sided [-12.12 to 2.42], Standard Error of Mean 3.56
Statistical Analysis 13: Comparison: Placebo vs PF-00489791 4 mg; mPAP at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.112, Longitudinal analysis; Adjusted Mean Difference = -6.01, 95% CI 2-sided [-13.51 to 1.49], Standard Error of Mean 3.67
Statistical Analysis 14: Comparison: Placebo vs PF-00489791 10 mg; mPAP at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.928, Longitudinal analysis; Adjusted Mean Difference = -0.34, 95% CI 2-sided [-7.91 to 7.23], Standard Error of Mean 3.71
Statistical Analysis 15: Comparison: Placebo vs PF-00489791 20 mg; mPAP at Hour 3: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.020, Longitudinal analysis; Adjusted Mean Difference = -9.01, 95% CI 2-sided [-16.52 to -1.50], Standard Error of Mean 3.68
Statistical Analysis 16: Comparison: Placebo vs PF-00489791 1 mg; mPAP at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.136, Longitudinal analysis; Adjusted Mean Difference = -5.80, 95% CI 2-sided [-13.55 to 1.94], Standard Error of Mean 3.79
Statistical Analysis 17: Comparison: Placebo vs PF-00489791 2 mg; mPAP at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.303, Longitudinal analysis; Adjusted Mean Difference = -3.82, 95% CI 2-sided [-11.27 to 3.63], Standard Error of Mean 3.65
Statistical Analysis 18: Comparison: Placebo vs PF-00489791 4 mg; mPAP at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.180, Longitudinal analysis; Adjusted Mean Difference = -5.17, 95% CI 2-sided [-12.87 to 2.52], Standard Error of Mean 3.77
Statistical Analysis 19: Comparison: Placebo vs PF-00489791 10 mg; mPAP at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.506, Longitudinal analysis; Adjusted Mean Difference = -2.56, 95% CI 2-sided [-10.31 to 5.20], Standard Error of Mean 3.80
Statistical Analysis 20: Comparison: Placebo vs PF-00489791 20 mg; mPAP at Hour 4: The analysis was performed using longitudinal analysis model with baseline as a covariate; Test type: Superiority or Other; p = 0.026, Longitudinal analysis; Adjusted Mean Difference = -8.84, 95% CI 2-sided [-16.54 to -1.14], Standard Error of Mean 3.77

8. Secondary Outcome: Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP), Mean Systemic Arterial Pressure (SAP), Systolic Systemic Arterial Pressure (sSAP) and Diastolic Systemic Arterial Pressure (dSAP) at Hour 1, 2, 3 and 4 Post Dose
Description: Hourly changes from baseline in hemodynamic parameters were reported. Hemodynamic parameters including PCWP, SAP, sSAP and dSAP were measured using a pressure transducer positioned at the mid-axillary line with the participant in the supine position. All hemodynamic pressure measurements (except PCWP for which 1 measurement is sufficient) were performed as triplicate measurements and average was used.
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6
mmHg
  Baseline: PCWP | 11.0 (1.79) | 8.2 (3.76) | 11.7 (1.70) | 7.3 (3.56) | 9.5 (2.07) | 10.4 (2.88) | 10.2 (1.72)
  Baseline: SAP: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  Baseline: SAP | 89.2 (14.06) | 91.0 (13.78) | 91.6 (11.62) | 96.0 (12.70) | 94.7 (10.69) | 95.5 (9.50) | 97.5 (10.58)
  Baseline: sSAP: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  Baseline: sSAP | 122.5 (12.76) | 132.0 (19.45) | 116.9 (6.07) | 131.2 (8.80) | 131.5 (15.67) | 126.5 (23.37) | 128.3 (15.81)
  Baseline: dSAP: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  Baseline: dSAP | 71.3 (12.55) | 67.0 (9.55) | 74.9 (12.81) | 77.2 (12.19) | 71.0 (8.46) | 78.2 (7.03) | 79.3 (7.00)
  PCWP: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 5
  PCWP: Change at hour 1 | -0.5 (2.43) | 0.3 (3.08) | -0.3 (0.49) | 0.8 (1.72) | 0.3 (1.37) | -1.7 (2.80) | -0.6 (1.52)
  SAP: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SAP: Change at hour 1 | -2.0 (7.13) | -5.8 (9.70) | -5.9 (7.93) | -6.3 (6.12) | -1.4 (6.36) | -6.7 (7.47) | -4.2 (6.08)
  sSAP: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  sSAP: Change at hour 1 | 2.3 (17.11) | -9.5 (16.28) | -0.6 (11.52) | -7.2 (5.64) | -2.3 (11.96) | -7.3 (8.16) | -5.2 (6.08)
  dSAP: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  dSAP: Change at hour 1 | -0.7 (1.63) | -4.3 (7.03) | -6.7 (8.96) | -5.0 (6.03) | -0.7 (4.23) | -7.2 (5.64) | -3.5 (5.82)
  PCWP: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 4 | 6 | 6 | 5
  PCWP: Change at hour 2 | 0.2 (2.48) | -0.3 (2.34) | -1.0 (1.15) | 0.0 (0.82) | -0.2 (1.33) | -1.7 (2.16) | -0.4 (1.14)
  SAP: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SAP: Change at hour 2 | -3.3 (7.03) | -6.1 (8.75) | -3.3 (10.00) | -5.3 (6.02) | -6.1 (11.44) | -6.8 (6.55) | -8.8 (10.07)
  sSAP: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  sSAP: Change at hour 2 | -0.5 (13.90) | -8.2 (14.93) | -0.7 (15.90) | -6.0 (4.90) | -5.2 (12.84) | -5.8 (9.66) | -10.3 (13.17)
  dSAP: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  dSAP: Change at hour 2 | -2.5 (4.46) | -4.3 (7.26) | -3.0 (9.87) | -3.0 (5.10) | -4.5 (8.19) | -7.7 (5.85) | -7.5 (8.09)
  PCWP: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 4 | 6 | 5 | 5
  PCWP: Change at hour 3 | -0.3 (2.07) | 0.8 (2.56) | -0.7 (1.11) | 0.3 (0.96) | 1.0 (4.00) | -0.8 (1.30) | -0.6 (1.52)
  SAP: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SAP: Change at hour 3 | -2.5 (9.20) | -1.5 (5.86) | -4.7 (9.09) | -7.0 (8.60) | -1.7 (22.10) | -10.5 (8.71) | -10.8 (12.09)
  sSAP: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  sSAP: Change at hour 3 | -0.3 (14.01) | -5.5 (11.15) | 1.3 (14.34) | -8.0 (10.66) | -9.2 (16.15) | -9.3 (13.75) | -12.2 (16.13)
  dSAP: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  dSAP: Change at hour 3 | -1.3 (5.82) | -1.2 (5.04) | -5.4 (8.70) | -6.7 (7.97) | -1.0 (15.03) | -9.5 (5.17) | -9.2 (10.30)
  PCWP: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 5 | 5
  PCWP: Change at hour 4 | -0.7 (1.51) | 0.8 (2.32) | -0.1 (1.35) | -0.7 (1.51) | 1.7 (3.78) | -1.0 (1.87) | 0.0 (0.00)
  SAP: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SAP: Change at hour 4 | -5.8 (9.02) | -4.3 (4.63) | -4.6 (7.63) | -4.3 (10.35) | -2.2 (8.08) | -9.0 (9.55) | -8.8 (11.86)
  sSAP: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  sSAP: Change at hour 4 | -1.3 (16.24) | -4.3 (9.69) | -1.7 (12.41) | -6.8 (13.63) | -4.7 (14.12) | -9.3 (15.13) | -10.8 (13.69)
  dSAP: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  dSAP: Change at hour 4 | -2.8 (7.36) | -2.3 (4.13) | -4.1 (8.05) | -3.7 (10.46) | -0.8 (6.11) | -7.7 (5.01) | -7.5 (10.88)

9. Secondary Outcome: Mean Change From Baseline in Pulmonary Vascular Resistance (PVR) and Systemic Vascular Resistance (SVR) at Hour 1, 2, 3 and 4 Post Dose
Description: Hourly changes from baseline in PVR and SVR were reported. PVR was calculated by: PVR (Wood units) = (mean PAP minus PCWP) divided by CO (taken as the average of the triplicate measurements). SVR (Wood units) = (mean SAP minus RAP) divided by CO (taken as the average of the triplicate measurements).
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Wood units
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6
Wood units
  PVR: Baseline | 1217.0 (765.98) | 665.1 (267.93) | 995.3 (638.42) | 1117.2 (523.04) | 820.5 (565.07) | 815.4 (600.27) | 966.6 (441.55)
  SVR: Baseline: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SVR: Baseline | 2122.7 (906.19) | 1537.4 (448.23) | 1648.8 (713.36) | 2089.7 (800.79) | 1873.9 (552.78) | 1654.8 (580.26) | 1948.8 (418.21)
  PVR: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 5
  PVR: Change at hour 1 | 60.2 (377.48) | -82.9 (158.83) | -24.2 (165.45) | -182.4 (306.17) | -147.1 (360.44) | -138.4 (85.91) | 67.9 (256.27)
  SVR: Change at hour 1: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SVR: Change at hour 1 | -125.0 (439.77) | -174.7 (231.65) | -139.0 (526.65) | -371.3 (678.24) | -373.1 (461.11) | -39.1 (128.88) | 63.9 (352.95)
  PVR: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 4 | 6 | 6 | 5
  PVR: Change at hour 2 | -19.8 (316.70) | -112.5 (129.43) | -6.5 (132.03) | -114.0 (487.12) | -196.7 (264.20) | -194.4 (207.82) | 142.8 (509.00)
  SVR: Change at hour 2: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SVR: Change at hour 2 | -281.4 (252.62) | -194.2 (296.66) | -173.7 (382.66) | -238.7 (715.18) | -538.9 (327.15) | -206.3 (208.43) | 12.7 (551.13)
  PVR: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 4 | 6 | 5 | 5
  PVR: Change at hour 3 | 0.9 (292.22) | -8.4 (112.08) | -3.2 (173.46) | -215.6 (549.52) | -153.9 (254.82) | -150.7 (272.64) | 223.3 (488.72)
  SVR: Change at hour 3: number analyzed (Participants) | 6 | 6 | 7 | 5 | 6 | 6 | 6
  SVR: Change at hour 3 | -269.3 (256.20) | -66.6 (189.66) | -93.8 (389.95) | -337.2 (935.47) | -432.3 (298.78) | -233.7 (272.19) | 30.9 (487.52)
  PVR: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 5 | 5
  PVR: Change at hour 4 | -28.9 (236.91) | -81.7 (127.73) | 10.5 (187.79) | -247.4 (281.78) | -188.5 (280.24) | -133.6 (219.26) | 260.9 (574.22)
  SVR: Change at hour 4: number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 6 | 6
  SVR: Change at hour 4 | -385.7 (290.25) | -53.2 (185.94) | -117.8 (412.25) | -505.2 (731.80) | -353.9 (403.12) | -215.6 (272.13) | 92.3 (517.94)

10. Secondary Outcome: Mean Change From Baseline in Heart Rate (HR) at Hour 1, 2, 3 and 4 Post Dose
Description: Hourly changes from baseline in HR were reported.
Time Frame: Baseline, 1, 2, 3, 4 hours post-dose on Day 1
Population: FAS included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6
beats per minute (bpm)
  Baseline | 78.2 (13.21) | 85.3 (16.28) | 90.1 (17.10) | 75.5 (14.05) | 77.2 (15.94) | 91.9 (17.90) | 86.7 (19.43)
  Change at hour 1 | -0.3 (11.60) | -3.5 (5.50) | -1.1 (5.01) | 4.3 (11.17) | 6.8 (7.31) | -0.9 (6.09) | -2.7 (6.47)
  Change at hour 2 | -0.5 (8.14) | -2.8 (3.60) | 0.1 (5.52) | 4.2 (9.37) | 9.7 (8.02) | -2.3 (4.75) | -0.5 (6.12)
  Change at hour 3 | -1.0 (10.39) | -1.2 (3.19) | -3.3 (9.66) | -1.8 (7.05) | 10.2 (4.12) | -3.1 (7.99) | -0.8 (6.82)
  Change at hour 4 | 1.5 (8.17) | -3.3 (2.80) | -2.0 (11.17) | 6.0 (8.34) | 5.7 (4.32) | -6.1 (6.72) | -0.5 (8.60)

11. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Criteria for clinically significant laboratory values:hemoglobin, hematocrit and red blood cells(less than[<]0.8*lower limit of normal[LLN]); leucocytes (<0.6*LLN/greater than[>]1.5*upper limit of normal[ULN]);platelets (<0.5*LLN></0>1.75* ULN);neutrophils, lymphocytes(<0.8*LLN></0>1.2* ULN); eosinophils, basophils, monocytes (>1.2*ULN);bilirubin (>1.5*ULN);aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase(>3*ULN);creatinine, blood urea nitrogen (>1.3*ULN);glucose(<0.6*LLN></0>1.5* ULN); uric acid(>1.2*ULN);sodium(<0.95*LLN></0>1.05*ULN); potassium, chloride, calcium(<0.9*LLN></0>1.1* ULN); albumin, total protein(<0.8></0>1.2* ULN); creatine kinase(>2.0*ULN);urine red blood cells(RBCs), urine white blood cells(WBCs)(>=6 per high-powered field);qualitative urine glucose, urine ketones, urine protein, urine blood/hemoglobin(>=1); urine bacteria(>20 per high-powered field); pregnancy test, urine protein, quantitative random serum pregnancy test (>=1).
Time Frame: Baseline up-to follow up (Day 3 to 5)
Population: Safety analysis set included all randomized participants who received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6
Participants | 3 | 3 | 3 | 3 | 3 | 3 | 3

12. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Values
Description: Criteria for clinically significant changes (changes of potential clinical concern) in ECG parameters: increase from baseline of >=30 to <60 milliseconds (msec) or >=60 msec in corrected QT interval (QTc), QT interval corrected using Fridericia's correction (QTcF) and QT interval corrected using Bazett's correction (QTcB); Increase from baseline of >= 25% (when baseline was >200 msec) or increase from baseline of >=50% (when baseline was <=200 msec) in PR interval; and Increase from baseline of >= 25% (when baseline was >100 msec) or increase from baseline of >=50% (when baseline was <=100 msec) in QRS interval. Number of participants with any clinically significant change in ECG values were reported.
Time Frame: Baseline up-to follow up (Day 3 to 5)
Population: Safety analysis set included all randomized participants who received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Mean Partial Pressure of Oxygen (PaO2) and Carbon Dioxide (PaCO2) at Hour 1 and 4 Post Dose
Description: Arterial blood samples for PaO2 and PaCO2 collected via an arterial line were assessed. PaO2 is the measure of oxygen level in the arterial blood and PaCO2 is the measure of carbon dioxide level in the arterial blood.
Time Frame: Baseline; 1, 4 hours post-dose on Day 1
Population: Safety analysis set included all randomized participants who received study medication. Here, N (overall number of participants analyzed) = participants evaluable for this measure and 'Number Analyzed' = participants who were evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 6 | 5 | 7 | 5 | 6 | 6 | 6
mmHg
  PaO2: Baseline | 64.1 (9.47) | 63.0 (14.92) | 65.4 (16.98) | 82.0 (16.32) | 72.4 (25.85) | 73.2 (15.75) | 64.9 (9.78)
  PaCO2: Baseline | 32.8 (4.79) | 32.0 (6.71) | 38.7 (7.53) | 31.4 (4.83) | 36.3 (6.09) | 39.3 (10.75) | 41.6 (15.07)
  PaO2: Change at Hour 1: number analyzed (Participants) | 6 | 5 | 7 | 5 | 5 | 5 | 6
  PaO2: Change at Hour 1 | -1.4 (11.06) | -4.4 (6.22) | -0.6 (7.98) | -6.5 (12.16) | -10.8 (12.99) | -13.7 (11.17) | 2.4 (12.48)
  PaCO2: Change at Hour 1: number analyzed (Participants) | 6 | 5 | 7 | 5 | 5 | 5 | 6
  PaCO2: Change at Hour 1 | 0.5 (2.69) | 1.4 (1.96) | -0.7 (3.70) | -0.2 (3.62) | -2.1 (2.98) | 1.4 (4.26) | -1.4 (3.77)
  PaO2: Change at Hour 4: number analyzed (Participants) | 6 | 5 | 7 | 5 | 5 | 6 | 6
  PaO2: Change at Hour 4 | 0.8 (8.03) | -0.4 (4.04) | 0.3 (13.47) | -4.0 (8.39) | -10.3 (9.65) | -7.7 (15.61) | 3.6 (7.47)
  PaCO2: Change at Hour 4: number analyzed (Participants) | 6 | 5 | 7 | 5 | 5 | 6 | 6
  PaCO2: Change at Hour 4 | -0.7 (1.36) | 1.0 (2.48) | -1.9 (4.44) | -1.6 (3.59) | -3.3 (2.91) | 0.6 (3.68) | 0.8 (10.55)

14. Secondary Outcome: Plasma Concentration of PF-00489791 and Sildenafil
Time Frame: 1, 2, 3, 4, 5, 6, 8 hours post-dose on Day 1, follow up (Day 3 to 5)
Population: Data was not reported for this outcome measure because the study was terminated and as per change in planned analysis, the pharmacokinetic parameters were not to be summarized.
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Safety population.
Arm/Group | Placebo | PF-00489791 1 mg | PF-00489791 2 mg | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20 mg | Sildenafil
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 0/7 | 0/6 | 0/6 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 2/7 | 5/6 | 4/6 | 2/7 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=6) | PF-00489791 1 mg (N=6) | PF-00489791 2 mg (N=7) | PF-00489791 4 mg (N=6) | PF-00489791 10 mg (N=6) | PF-00489791 20 mg (N=7) | Sildenafil (N=6)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5 | 0/5 | 0/4 | 0/4 | 0/3 | 1/5 | 0/4 — This was a gender specific event.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | PF-00489791 1 mg (N=6) | PF-00489791 2 mg (N=7) | PF-00489791 4 mg (N=6) | PF-00489791 10 mg (N=6) | PF-00489791 20 mg (N=7) | Sildenafil (N=6)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary sediment present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated prematurely as further continuation would not have meaningfully contributed to the next phase of development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.